CLINICAL TRIAL: NCT01196910
Title: Test Efficiency of Deep Transcranial Magnetic Stimulation (DTMS) Using an H-coil for Dorso-Lateral Prefrontal Cortex (HLPFC) to Treat Attention Deficit Hyperactivity Disorder (ADHD) in Adults
Brief Title: Deep Transcranial Magnetic Stimulation (DTMS) as a Treatment for Attention Deficit Hyperactivity Disorder (ADHD) in Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBR-0014-00
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stimulation over the left dorsolateral prefrontal cortex (Active Comparator): Group A (fifteen subjects) - treatment by HLPFC coil high-frequency stimulation over the left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: treatment by HLPFC coil
- stimulation over the right DLPFC (Active Comparator): Group B (fifteen subjects) - Treatment by HLPFC coil high-frequency stimulation over the right DLPFC.
  Interventions: Device: treatment by HLPFC coil
- Treatment with HLPFC coil simulator mode (Placebo Comparator): Group C (fifteen subjects) - Treatment with HLPFC coil simulator mode (sham).
  Interventions: Device: treatment by HLPFC coil

INTERVENTIONS:
Device: treatment by HLPFC coil — DTMS treatment will be given for 3 weeks, 5 days a week. Before each DTMS treatment, neural network excitation practice will be done using AttenGo software (AttenGo, Herzlia, Israel).
  Each treatment day: Follow-up to evaluate clinical side effects of treatment. Two additional meetings with DTMS treatment and follow-up will be held to evaluate the efficacy of treatment and side effects. The first will be four weeks after the end of the daily treatment phase; the second eight weeks after the end of the daily treatment phase.

SUMMARY:
The aim of the study is to assess the effect of left or right high-frequency DTMS on ADHD symptoms, cognitive performance and decision-making ability of ADHD adults, and to compare this to the effect of sham DTMS on ADHD adults

DETAILED DESCRIPTION:
Attention deficit disorder in adults may be due to hypoactivity of prefrontal areas of the brain. Increasing the activity of these areas may help improve symptoms in many of these patients. In addition there is evidence as to dysfunction in both hemispheres of the brain, but it is difficult to determine the contribution of each hemisphere's pattern of activity to behavioral impairment. The purpose of this study is to use high-frequency DTMS to stimulate activity either on the left side of the prefrontal cortex (one arm), or on the right side (a second arm), to see if such stimulation improves attention, comparing to sham DTMS simulation (a third arm).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-65.
* Appropriate diagnosis of ADHD according to DSM-IV criteria:

  o DSM-IV criteria require not only that the ADHD symptoms be present now (self-report), but also to have been present in childhood (self-report)
* Subjects taking medications for attention deficit disorder will give their consent to stop the drugs from a week before the start of participation in the study, and during the daily treatment phase (four weeks total); subjects also will be asked not to take these medications 24 hours before participation in the review meetings (4 and 8 weeks after the end of the daily treatment phase).
* Subjects have given their written and oral consent to participate in research.

Exclusion Criteria:

* Any DSM-IV Axis I psychiatric disorder.
* Use of antipsychotic stabilizers; other than benzodiazepines if necessary to a daily dosage equivalent to 2 mg Lorazepam.
* History of lack of tolerance to TMS.
* Diagnosis of severe DSM-IV personality disorder.
* Current suicidal tendency.
* Uncontrolled high blood pressure
* History of epilepsy, seizures or fever convulsions.
* History of epilepsy or convulsions in first-degree relatives.
* A history of head injury or a stroke which caused deficits.
* History of metal in the head (outside the oral cavity).
* History of plastic or metal implants, including metallic particles in the eye, pacemaker, implanted hearing aid devices, use of neurostimulators, or any medical pump.
* A history of drug or alcohol misuse.
* People who lack judgment or are unable to communicate with the experimenters.
* Participation in any other medical research during the three months prior to the time of this experiment.
* Subject's inability to sign a consent form.
* Pregnancy, or not using contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-07; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Conners' Adult ADHD Rating Scale | Screening, at the end of three weeks of treatment, and for each of two follow-up meetings

SECONDARY OUTCOMES:
Mindstreams Cognitive Tests | Screening, at the end of three weeks of treatment, and for each of two follow-up meetings

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Bleich-Cohen M, Gurevitch G, Carmi N, Medvedovsky M, Bregman N, Nevler N, Elman K, Ginou A, Zangen A, Ash EL. A functional magnetic resonance imaging investigation of prefrontal cortex deep transcranial magnetic stimulation efficacy in adults with attention deficit/hyperactive disorder: A double blind, randomized clinical trial. Neuroimage Clin. 2021;30:102670. doi: 10.1016/j.nicl.2021.102670. Epub 2021 Apr 18. PMID 34215144